CLINICAL TRIAL: NCT06354946
Title: External Validation of Simplified 4C Mortality Score by Deleting CRP
Acronym: 4Cs
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, PROFESSOR, University of Monastir
Other Study IDs: SCORE 4C
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: COVID-19 Pandemic
Keywords: SCORE 4C; SARS-COV2; validation; deleting CRP
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The (Coronavirus Clinical Characterisation Consortoum) 4C mortality score is an accessible risk stratification score developed by the International Severe Acute Respiratory and Emerging Infections Consortium (ISARIC) based on eight different parameters: age, sex, number of comorbidities, respiratory rate, peripheral oxygen saturation, level of consciousness (Glasgow Coma Scale), urea or blood urea nitrogen (BUN) level, and C reactive protein (CRP). It was derived and internally validated on a large, diverse cohort within the United Kingdom but requires external validity to confirm its generalizability. A recent validation study demonstrated that the score could be simplified by deleting CRP item which is favorable to its widespread use. we aim to validate a modified 4C score.

DETAILED DESCRIPTION:
The clinical presentation and progression of COVID-19 in patients is highly variable, which makes it difficult for clinicians to triage patients and determine their prognostic risk.

The (Coronavirus Clinical Characterisation Consortoum) 4C mortality score is an accessible risk stratification score developed by the International Severe Acute Respiratory and Emerging Infections Consortium (ISARIC) based on eight different parameters: age, sex, number of comorbidities, respiratory rate, peripheral oxygen saturation, level of consciousness (Glasgow Coma Scale), urea or blood urea nitrogen (BUN) level, and C reactive protein (CRP). It was derived and internally validated on a large, diverse cohort within the United Kingdom but requires external validity to confirm its generalizability. A recent validation study demonstrated that the score could be simplified by deleting CRP item which is favorable to its widespread use. The study aim to validate a modified 4C score.

Methods

This is a multicenter retrospective observational, cohort study of patients admitted to five Tunisian university hospitals (Fattouma Bourguiba Hospital Monastir, Sahloul Hospital Sousse, Farhat Hached Hospital Sousse, Taher Sfar Hospital Mahdia, Habib Bourguiba Hospital Sfax, Traumatology and Burns Center Tunis), the study included medical records of all adult patients with confirmed COVID-19 infection who were hospitalized from January 2020 and November 2022. A confirmed case of COVID-19 was defined by a positive reverse transcriptase-PCR (RT-PCR) assay of a nasopharyngeal swab associated with compatible clinical manifestations. Incomplete electronic record were excluded from the analysis.

Anamnesis, clinical, paraclinical, radiological, and outcome data were collected using a validated electronic case report form (eCRF). The primary outcomes measure was in-hospital death from any cause.

ELIGIBILITY:
Inclusion Criteria:

- admitted to one of the participating hospitals with a confirmed case of COVID-19 defined by a positive reverse transcriptase-PCR (RT-PCR) assay of a nasopharyngeal swab associated with compatible clinical manifestations

Exclusion Criteria:

* Incomplete electronic records were excluded from the analysis.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a multicenter retrospective observational, cohort study of patients admitted to five Tunisian university hospitals (Fattouma Bourguiba Hospital Monastir, Sahloul Hospital Sousse, Farhat Hached Hospital Sousse, Taher Sfar Hospital Mahdia, Habib Bourguiba Hospital Sfax, Traumatology and Burns Center Tunis), the study included medical records of all adult patients with confirmed COVID-19 infection who were hospitalized from January 2020 and November 2022. A confirmed case of COVID-19 was defined by a positive reverse transcriptase-PCR (RT-PCR) assay of a nasopharyngeal swab associated with compatible clinical manifestations. Incomplete electronic record were excluded from the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome was all-cause in-hospital mortality rate The primary outcome was all-cause in-hospital mortality rate | 30 days after inclusion
  The primary outcomes measure was in-hospital death from any cause.

SECONDARY OUTCOMES:
Number of patients admitted to the ICU | 30 days after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Khaoula Bel Haj Ali, Principal Investigator — CHU Fattouma Bourguiba Monastir, service des urgences
Locations (1):
- EPS Fattouma Bourguiba University hospital, Monastir, Tunisia